CLINICAL TRIAL: NCT02899741
Title: Efficacy of Omega-3 as Adjunctive Therapy for Medically Intractable Epilepsy: A Prospective Open-label Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508174702
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Epilepsy
Keywords: Medically intractable epilepsy, Omega-3
MeSH Terms: conditions — Epilepsy | interventions — Docosahexaenoic Acids; Omacor

ARMS (1):
- Omega-3 (Experimental): One group of this study. Omega-3 will be administered for thee months.
  Interventions: Drug: Omega-3

INTERVENTIONS:
Drug: Omega-3 — 1000mg every day for 90 days
  Other Names: Omega-3, Omacor

SUMMARY:
The purpose of this study is to determine whether omega-3 is effective in the treatment of medically intractable epilepsy as adjunctive therapy.

DETAILED DESCRIPTION:
This study will enroll total 30 patients with medically intractable epilepsy. The patients will be fully assessed on the enrollment, and then seizure frequency will be counted for three months without changing medication. After three months, Omega-3 will be administered for next three months. Seizure frequency, questionnaires evaluating mood and QOL, and adverse events are evaluated at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medically intractable, focal or generalized, epilepsy: Patients with localization-related partial onset or generalized tonic/clonic seizure according to the International League Against Epilepsy (ILAE) can be included. Medically intractable epilepsy means that recurrent seizures occur even though two or more anti-epileptic drugs have been used appropriately for over one year.
* Seizure frequency criteria: three seizures per one month for recent 3 months before enrollment
* Seizure criteria: simple partial, complex partial, or tonic-clonic seizures
* Subjects with normal cognitive function: patients who can perform normal daily life. If not definite, enrollment will be done with K-MMSE score over 27.

Exclusion Criteria:

* Poor general medical condition: comorbid with heart, lung, liver diseases
* Patients who have history of pseudo-seizure
* Anti-epileptic drugs has been changed in recent one month.
* Chronic alcoholic
* Seizure count cannot be done since seizures occur successively.
* Allergy to fish
* High risk of bleeding such as trauma or operation
* Liver function abnormality
* Pregnant or lactating women, or women who plans to have children
* Patients who have participated in the other clinical trial in recent one month

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | three months

SECONDARY OUTCOMES:
Depressive mood | three months
  BDI-2 questionnaire
Anxiety | three months
  HAM-A questionnaire
Quality of Life | three months
  SF-36 v2 questionnaire
Adverse events | three months

CONTACTS AND LOCATIONS:
Overall Officials: Kon Chu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No